CLINICAL TRIAL: NCT02661191
Title: Effect of Vitamin D Repletion on Asthma Exacerbation
Brief Title: Vitamin D Deficiency and Asthma Exacerbation
Acronym: AVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Caterina Bucca, Professor of Respiratory Medicine, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTHMAVITD
Record Dates: First submitted 2015-12-21; First posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Asthma; Vitamin D Deficiency; Disease Exacerbation
Keywords: asthma; vitamin D; exacerbations; airway obstruction
MeSH Terms: conditions — Asthma; Vitamin D Deficiency; Disease Progression; Airway Obstruction | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- asthma severity and disease exacerbation (Other): intramuscular cholecalciferol 100,000 IU, followed by oral cholecalciferol 5000 IU weekly plus 400 IU daily for one year
  Interventions: Drug: oral cholecalciferol

INTERVENTIONS:
Drug: oral cholecalciferol — Inhaled corticosteroids and long-acting beta-agonists, salbutamol
  Other Names: intramuscular cholecalciferol

SUMMARY:
The study aim is in two phases. First phase: to evaluate the influence of vitamin D deficiency on asthma severity, degree of airway obstruction and frequency of asthma exacerbations. Second phase: to evaluate if in patients with vitamin D deficiency (25-OH vitamin D levels below 20 ng/ml), vitamin D supplementation decreases the number of disease exacerbations.

DETAILED DESCRIPTION:
The first phase of the study consisted of a cross-sectional examination of a cohort of 119 asthmatic patients, who had at least one year regular follow-up in our respiratory clinic, and were not receiving any vitamin D supplementation.

In the second phase patients with vitamin D deficiency (25-OH D values below 20 ng/ml), were recruited in a one year longitudinal study, during which they received vitamin D supplementation. The study started and ended in late autumn-winter season when, at our latitude, sun exposure is lowest. Symptoms, spirometry and number of exacerbations were recorded during both study phases.

ELIGIBILITY:
Inclusion Criteria:

* All the consecutive patients with bronchial asthma of any severity, who presented for a scheduled visit at our Respiratory Clinic during the period October 2012-March 2013 and who had at least one year regular follow-up every three months

Exclusion Criteria:

* Acute exacerbation in the last month and treatment with vitamins and dietary supplements in the last year.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Relationship between serum 25-hydroxide (OH) vitamin D level and asthma exacerbations (number/year= unscheduled visits for worsening symptoms, increase in therapy) | one year
  119 consecutive asthmatic patients underwent serum vitamin D (25-OHD) and lung function assessment. Their medical records were retrospectively reviewed, to gain information on disease exacerbations during the 12 months preceding study entry. The relationship between baseline 25-OH vitamin D and number of exacerbation was investigated
Effect of vitamin D supplementation in patients with 25-OH vitamin D < 20 ng/ml on asthma exacerbations (number/year= unscheduled visits for worsening symptoms, increase in therapy) | One year
  55 asthmatic patients with 25-OH vitamin D below 20 ng/ml underwent supplementation with cholecalciferol for one year (intramuscular 100,000 IU, followed by oral 5000 IU weekly plus 400 IU daily for one year). Number of exacerbations were recorded during the year of supplementation and compared with the data recorded during vitamin D deficiency

SECONDARY OUTCOMES:
Relationship between serum 25-OH vitamin D level and airway obstruction (evaluated by spirometry: one second forced expiratory volume, FEV1 l/sec, vital capacity (VC) and FEV1/VC%) | one year
  119 consecutive asthmatic patients underwent serum vitamin D (25-OHD, ng/ml) and lung function assessment. Their medical records were retrospectively reviewed, to gain information on lung function tests (forced expiratory volume in 1 second, FEV1, and vital capacity, VC) during the 12 months preceding study entry. The relationship between baseline 25-OH vitamin D and airway obstruction (FEV1 and FEV1/VC%) was investigated
Effect of vitamin D supplementation in patients with 25-OH vitamin D < 20 ng/ml on airway obstruction ( FEV1 l/sec, FEV1/VC%) | one year
  55 asthmatic patients with 25-OH vitamin D below 20 ng/ml underwent supplementation with cholecalciferol for one year (intramuscular 100,000 IU, followed by oral 5000 IU weekly plus 400 IU daily for one year). Lung function tests (FEV1, VC and FEV1/VC%) were recorded during the year of supplementation and compared with the data recorded during vitamin D deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Caterina B Bucca, MD, Study Chair — Dept. Medical Science, University of Turin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malinovschi A, Masoero M, Bellocchia M, Ciuffreda A, Solidoro P, Mattei A, Mercante L, Heffler E, Rolla G, Bucca C. Severe vitamin D deficiency is associated with frequent exacerbations and hospitalization in COPD patients. Respir Res. 2014 Dec 13;15(1):131. doi: 10.1186/s12931-014-0131-0. PMID 25496239
- [Background] Masoero M, Bellocchia M, Ciuffreda A, Ricciardolo FL, Rolla G, Bucca C. Laryngeal spasm mimicking asthma and vitamin d deficiency. Allergy Asthma Immunol Res. 2014 May;6(3):267-9. doi: 10.4168/aair.2014.6.3.267. Epub 2014 Jan 14. PMID 24843804